CLINICAL TRIAL: NCT06257225
Title: Radiographic And Clinical Evaluation of Horizontal Bone Gain in the Lower Posterior Partially Edentulous Patients Comparing the Stabilization of The Resorbable Collagen Membrane With and Without Tacs
Brief Title: Evaluation of Horizontal Bone Gain in the Lower Posterior Partially Edentulous Patient Comparing the Stabilization of Membranes With and Without Tacs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Misr International University (Other)
Responsible Party: Principal Investigator, Hani Elnahass, Professor of Periodontology, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PerioMIU1029
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Guided Bone Regeneration
Keywords: GBR; Tacs
MeSH Terms: conditions — Spondylocostal Dysostosis 4, Autosomal Dominant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient showing horizontal defect and treated with GBR stabilized with Tacs (Active Comparator): Fixation
  Interventions: Procedure: Guided Bone regeneration
- Patient showing horizontal defect and treated with GBR stabilized with no Tacs (Experimental): No Fixation
  Interventions: Procedure: Guided Bone regeneration

INTERVENTIONS:
Procedure: Guided Bone regeneration — After local anesthesia, a crestal incision will be performed followed by full-thickness mucoperiosteal flap elevation Flap advancement will be attained through periosteal scoring of the buccal; The resorbable collagen membrane (Bio Gide, Geistlich AG) will be trimmed to the defect size. Xenograft (Bio-Oss) together with scrapped autogenous bone will be mixed and placed at the surgical site. The membrane will positioned over the graft and tucked into the lingual flap. Patient allocation concealment will be broken and the patients will be randomly assigned into two groups Patients receiving horizontal bone augmentation with resorbable collagen membrane stabilized with no tacks. The first layer will be closed with horizontal mattress sutures placed 4 mm from the incision line, and single interrupted sutures are used to close the edges of the flap. Vertical incisions are closed using single interrupted sutures and mattress suture should remain in place for at least 2 to 3 weeks

SUMMARY:
To address the gap of knowledge in comparing between the bone augmentation outcomes with or without tacks for membrane stabilization

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least 1 missing tooth in the posterior mandibular area Patients with an age above 18 years Systemically healthy patients

Healed alveolar ridge for implant placement with:

* Deficient buccolingual dimension ( ≤5mm)
* Sufficient vertical height (≥ 10 mm)
* Sufficient mesio-distal width (≥ 6.5 mm) Inter-arch space ≥ 7 mm to allow space for implant-supported crown Presence of neighboring and opposing dentition Soft tissue phenotype with keratinized tissue width (KTW) (≥2 mm) and gingival thickness (≥2 mm) Good oral hygiene Cooperative patients who accepted the trial follow up period and sign the informed consen

Exclusion Criteria:

* Systemic diseases or medications that might affect bone metabolism, increase surgical risk or complicate post-operative healing Untreated periodontal diseases History of radiation therapy to the head and neck Heavy smokers (≥ 10 cigarettes per day) Pregnant or lactating females Alcoholism or drug abuse Psychiatric problems Patients with signs of acute infection related to the area of interest

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Horizontal bone gain assessed radiographically (mm) | Baseline , 4 month
  Using CBCT

SECONDARY OUTCOMES:
Horizontal bone gain assessed clinically (mm) | Baseline , 4 month
  Bone Caliper
Amount of Pain | 7 days
  Visual Analogue Scale (VAS) (Price et al., 1983)
Amount of Pain | 7 days
  Number of analgesics consumed daily for 7 days
Patient satisfaction | 4 month
  Questionnaire - Binary
Surgical Time | During Surgery
  Stop Watch
Histological Evaluation | 4 month
  Core Biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Hani ElNahass, PhD, Principal Investigator — Cairo University; Omnia Tawfik, PhD, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided
I will check with Study chair